CLINICAL TRIAL: NCT05766566
Title: Treatment of Perianal Fistulas in Crohn's Disease With Autologous Microfragmented Adipose Tissue With the Lipogems® System
Brief Title: Treatment of Perianal Fistulas in Crohn's Disease With Autologous Microfragmented Adipose Tissue With the Lipogems System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Dr. Fabio Marino - MD, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: Lipogems
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Crohn Disease; Fistula; Adipose Tissue
Keywords: Lipogems
MeSH Terms: conditions — Crohn Disease; Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Will be enrolled patients referring to the Department of General Surgery of the IRCCS "Saverio de Bellis" - Castellana Grotte (BA) Italy, affected by perianal fistulas from Crohn's disease.
  Interventions: Procedure: Perianal fistula surgery

INTERVENTIONS:
Procedure: Perianal fistula surgery — surgical treatment of the perianal fistula through curettage, closure with suture thread (vicryl 2/0) of the internal orifice and lipofilling of the passage with microfragmented autologous adipose tissue processed with the Lipogems® system.

SUMMARY:
The aim of the study is to verify the efficacy of microfragmented autologous adipose tissue with the Lipogems® system, in the treatment of perianal fistulas of m. Crohn's.

The Lipogems® International, Milan, Italy, system is a sterile and disposable device that allows to harvest adipose tissue, process it and use it for intraoperative autologous transplantation of human adipose tissue mesenchymal cells that have a gene expression profile and phenotypic similar to that of adipose stem cells.

The system consists of a container with metal beads capable of carrying out, by handling, a mechanical micro-fragmentation of the lipoaspirate and of a washing and filtering system which allows to progressively reduce the size of the adipose tissue clusters down to 0.2-0.8 mm and eliminate blood and oily residues.

The processed Lipogems® is fluid and easily injectable and is rich in mesenchymal cells and pericytes.

The processed Lipogems® will be injected around the fistulous tract and the tissue area closing the internal orifice to promote healing.

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory disease of unknown etiology, probably multifactorial, which can affect the entire digestive tract but especially the terminal ileum. Its incidence is increasing exponentially, resulting in a growing care commitment and an increasingly onerous economic burden for the NHS.

In 25% - 80% of patients with m. Crohn's disease there is an involvement of the perianal tissues due to particularly disabling symptoms such as pain, chronic mucopurulent secretions, recurrent acute septic episodes which, in over a third of cases, result in complex anal and ano-vaginal fistulas with the need for hospitalization multiple and significant impairment of the quality of socio-relational and working life.

The treatments currently available for perianal Crohn's are mainly based on the use of biological drugs known both for their high cost and for their important side effects, but 37% of patients present recurrence or persistence of the disease with the need to resort to surgery . In about 90% of cases, the surgery is repeated more than once, resulting in a significantly increased risk of faecal incontinence.

Sometimes a stoma and proctectomy may be necessary. Göttgens KW et al. highlight how, in the last twenty years, the risk of developing a perianal fistula has remained substantially stable, as well as its recurrence rate, underlining the need to improve treatment strategies.

The COVID-19 pandemic has further complicated the clinical management of patients with m. Crohn's disease both due to the need to limit their mobility and access to healthcare settings and due to the fear that immunosuppressive and immunomodulatory therapies could expose them to a greater risk of infection and complications. Although an increase in the incidence of SARS COVID-19 infection is not currently demonstrated in this subpopulation of patients, it could, however, be more vulnerable to COVID-19. In fact, it has been seen how the SARS-CoV 2 virus enters the cells by binding to the ACE2 receptors which are overexpressed at the level of the inflamed intestinal epithelium and constitute a potential entry route for the virus into the human body. Furthermore, a recent international survey has shown that it is common practice to suspend biological therapy in patients with m. Crohn's disease infected with SARS-CoV 2.

In sight of these premises, it appears necessary to direct scientific research towards the study of alternative treatments that can prove to be more effective and safer in the treatment of perianal Crohn's.

Some authors have hypothesized that the high rate of failure in healing of perianal fistulas may be related to the poor tissue repair capacity that patients with m. Crohn's. Scientific studies have shown that adult stem cells isolated from adipose tissue have the possibility of differentiating into different histotypes including specialized muscle cells. Other studies have seen that in the aspirate of human adipose cells there is a pool of pluripotent mesenchymal stem cells that can differentiate into both myocytes and adipocytes and chondrocytes. Finally, it has been seen that stem cells isolated from human adipose tissue have the property of regulating the immune response through the production/modulation of a cytokine storm. In fact, some researchers have demonstrated that the systemic intravenous administration of stem cells taken from human adipose tissue can improve the clinical conditions of experimental mouse models in which both colitis and a septic state had been induced. Mesenchymal stem cells appear to act by migrating towards inflamed sites, promoting the secretion of molecules with an anti-inflammatory action such as IL10, IL 6, HGF, TGFB1 and indolamine 2,3 dioxygenase and, through a further paracrine action which locally maintains the anti-inflammatory effect . It has also been seen how mesenchymal stem cells are able to promote the action of CD4+ T lymphocytes which are notoriously deficient in m. Crohn's. Finally, the immunomodulatory activity of mesenchymal stem cells appears to influence the activity of dendritic cells and macrophages as well as lymphocytes.

Allogeneic adipose mesenchymal stem cells appear to be well tolerated by patients who receive them not expressing class II HLA antigens.

Adipose stem cells, compared to mesenchymal stem cells taken from the bone marrow, seem to replicate faster and for longer in culture and, moreover, they seem to produce higher levels of immunomodulatory cytokines such as IL6 and TGFB1.

The Lipogems® system is a sterile and disposable device that allows to harvest adipose tissue, process it and use it for intraoperative autologous transplantation of human adipose tissue mesenchymal cells that have a gene expression and phenotypic profile similar to that of adipose stem cells. The entire procedure takes place in a single surgical stage, in a closed circuit and with minimal tissue manipulation. The system consists of a container with metal beads capable of carrying out, by handling, a mechanical micro-fragmentation of the lipoaspirate and of a washing and filtering system which allows to progressively reduce the size of the adipose tissue clusters down to 0.2-0.8 mm and eliminate blood and oily residues. The processed Lipogems® is fluid and easily injectable and is rich in mesenchymal cells (in quantities 2-3 times greater than the classic lipoaspirate) and pericytes. Furthermore, the preservation of a stromal niche architecture increases cell viability and improves the cellular ability to respond to the stimuli of a regenerating environment. The processed Lipogems® will be injected around the fistulous tract and the tissue area closing the internal orifice to promote healing. Some studies have been published which, although on a limited number of patients with Crohn's fistulas, show a curative potential of Lipogems®. The literature, however, requires both prospective studies and studies on an adequately large sample of patients. Furthermore, there are no assessments relating to the quality of life of patients treated with Lipogems®.

The study involves three phases:

1. SCREENING: a first phase of patient selection by means of a pelvic-perianal MRI study and discussion of the clinical case with the dedicated gastroenterologist (patients with single channel or prevalent fistulous channel will be included who are non-responders to medical and/or seton therapy). In this phase there will also be a baseline assessment of the quality of life with the Crohn's Anal Fistula Quality of Life (CAF-QoL) score.
2. A second operative phase of surgical treatment of the perianal fistula through curettage, closure with suture thread (vicryl 2/0) of the internal orifice and lipofilling of the passage with microfragmented autologous adipose tissue processed with the Lipogems® system.
3. A third phase of follow-up lasting at least 2 months to evaluate whether or not the fistula was clinically healed (no discomfort, absence of secretions from the external orifice, reassessment of quality of life with the CAF-QoL) and any complications .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 and under 80 of both sexes
* Patients with single or multiple perianal fistulae of M. Crohn's not amenable to fistulotomy(due to involvement of the sphincters)
* Patients without acute local sepsis
* Patients who have had Crohn's disease in stable remission for at least 6 months.
* Previously treated patients (recurring fistulas) will also be included. Even the presence of a stoma or lax seton will not constitute grounds for exclusion.

Exclusion Criteria:

* Patients with cryptogenic perianal fistulas
* Patients with large incisional hernias that could favor intestinal perforations during the abdominal liposuction phase
* Patients with history of previous neoplastic pathologie

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to the Department of General Surgery of the IRCCS "Saverio de Bellis" - Castellana Grotte (BA) Italy, affected by perianal fistulas from Crohn's disease will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Demonstration of fistula healing | Two months after surgery
  Demonstration of fistula healing by proctological objective examination.

SECONDARY OUTCOMES:
Positive change in quality of life | Evaluation at screening and follow-up, two months after surgery
  Demonstrate a positive change in the quality of life of treated patients by administering the questionnaire: Crohn's Anal Fistula Quality of Life (CAF-QoL) score.
  The score of this questionnaire ranges between 0 and 112. The higher score indicates the worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Marino, MD, Principal Investigator — IRCCS "Saverio de Bellis" - Castellana Grotte (BA) - Italy
Locations (1):
- Unit of General Surgery, National Institute of Gastroenterology - IRCCS "Saverio de Bellis", Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruffolo C, Citton M, Scarpa M, Angriman I, Massani M, Caratozzolo E, Bassi N. Perianal Crohn's disease: is there something new? World J Gastroenterol. 2011 Apr 21;17(15):1939-46. doi: 10.3748/wjg.v17.i15.1939. PMID 21528071
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Rius J, Nessim A, Nogueras JJ, Wexner SD. Gracilis transposition in complicated perianal fistula and unhealed perineal wounds in Crohn's disease. Eur J Surg. 2000 Mar;166(3):218-22. doi: 10.1080/110241500750009311. PMID 10755336
- [Background] Mizuno H, Zuk PA, Zhu M, Lorenz HP, Benhaim P, Hedrick MH. Myogenic differentiation by human processed lipoaspirate cells. Plast Reconstr Surg. 2002 Jan;109(1):199-209; discussion 210-1. doi: 10.1097/00006534-200201000-00030. PMID 11786812
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456